CLINICAL TRIAL: NCT05419557
Title: Buen Provecho!: A Virtual Family-Based Intervention to Promote Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U21-12-4630
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-07

CONDITIONS: Health Behavior; Diet, Healthy; Childhood Obesity
MeSH Terms: conditions — Health Behavior; Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: concurrent groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): 12 week virtual family-based health eating program
  Interventions: Behavioral: Virtual Family-Based Healthy Plate Club
- Comparison (No Intervention): Standard in-office counseling about diet

INTERVENTIONS:
Behavioral: Virtual Family-Based Healthy Plate Club — IHPC provides produce boxes, nutrition and meal-preparation, education, and supportive counseling to address barriers related to obtaining produce and food. The intervention provides participants with a bi-weekly produce box for 12 weeks and helps families identify sustainable ways to obtain vegetables once the produce boxes end. The CHW will support families by coaching them on how to prepare these unfamiliar vegetables, give tips on finding sales at grocery stores, as well as by navigation to food assistance sites including food pantries. Parents will learn strategies to increase vegetable consumption by addressing perceived barriers - such as the child doesn't like vegetables. Curriculum will also include topics such as how to increase physical activity and reduce screen time.
  Arms: Intervention

SUMMARY:
The purpose of this pilot study is to compare the effectiveness of an expanded virtual educational program at modifying knowledge, self-efficacy, and behaviors when compared to traditional in-office counseling for guardians of children who are obese or overweight.

DETAILED DESCRIPTION:
Rationale: Obesity rates are significantly higher among Hispanic youth in the United States, disproportionately putting these children at an increased risk for obesity-related diseases such as hypertension, dyslipidemia, and impaired glucose tolerance. While virtual programming offers an innovative option for pediatric weight management, limited data exists on the efficacy of virtual interventions for this population and their guardians (parents / caregivers).

Objectives: The purpose of this pilot study is to compare the effectiveness of an expanded virtual educational program (expanded -Inova Healthy Plate Club, x-IHPC) at modifying knowledge, self-efficacy, and behaviors when compared to traditional in-office counseling for guardians of children who are obese or overweight.

Study Design: In order to test the effectiveness of the x-IHPC intervention, outcomes from participants in this pilot study will be compared with outcomes from a comparison group of similar participants who receive standard nutrition counseling during their regularly scheduled check-ups. The team will enroll 25 children in the x-IHPC intervention and the same number in the comparison group (n=50). Both groups will receive standard in-office counseling, but the intervention group will also receive the x-IHPC.

Study Methodology: The comparison group receives standard, in-office counseling at visits 1, 3-months and 6-months. The intervention group receives standard in-office counseling at the same intervals, and also participates in a 12-week x-IHPC developed by a dietician curriculum specialist. In addition, a key pillar of this study is identifying and training Community Health Workers (CHWs) to be Spanish-speaking facilitators of the x-IHPC and utilizing community engagement strategies. Training these CHWs and including them in designing the x-IHPC curriculum, will ensure that the programming is culturally appropriate; includes local features that relate directly to the community's needs; and enables study facilitators to respond effectively to the questions and learning needs of the parents and children involved in the program.

Statistical Methodology:

To examine the research question, a longitudinal analysis using generalized estimating equations (GEE) will be conducted to assess if mean differences exist on dietary measures, screen time, sleep quality, physical activity and guardian self-efficacy and confidence between the intervention and comparison groups while accounting for the correlation among the repeated measurements and controlling for covariates.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria include:

1. Child is clients at community clinic
2. Child between the ages 6-12 years
3. Child has a BMI percentage greater than 85%
4. Primary parent or guardian is > 18 years of age
5. Family identifies as Hispanic and Spanish is one of the primary languages spoken in the home
6. Children will be living with the primary guardian or parent for the duration of the program
7. Access to the internet
8. Parent or guardian is willing to commit to engaging in the 12 week program

Exclusion Criteria:

1. Family plans to change location within the year
2. During initial screening for the study, the study PI determines that the intervention may exacerbate existing medical conditions of the child or the family.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- HealthWorks for Northern Virginia, Leesburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Occurred between 08/18/2022 and 10/10/2022
Pre-assignment Details: None. All participants enrolled were assigned to a group.
Period: Overall Study
Arm/Group | Intervention | Comparison
Started | 22 | 20
Completed | 11 | 16
Not Completed | 11 | 4
Not completed — Lost to Follow-up | 11 | 4

BASELINE CHARACTERISTICS:
Groups:
- Comparison: Standard in-office counseling about diet, physical activity and screen time
- Total: Total of all reporting groups
Arm/Group | Intervention | Comparison | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 20 | 42
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 12 Withdrew from the study, 3 lost to Follow-Up
  Participants
    number analyzed (Participants) | 11 | 16 | 27
    Hispanic or Latino | 10 | 14 | 24
    Not Hispanic or Latino | 1 | 2 | 3
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 12 Withdrew, 3 Lost to Follow-Up
  Participants
    number analyzed (Participants) | 11 | 16 | 27
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 11 | 15 | 26
    More than one race | 0 | 1 | 1
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants Who Consumed Vegetables With Their Dinner Meal More Than 5 Days Per Week
Description: Days per week child ate vegetables with dinner meal, post intervention Measured with a food frequency questionnaire, question: "Think about all the foods your child ate at your dinner/supper meal and snacks in the past week. On how many days did your child eat vegetables for the dinner meal?" Answer options: 1, Never | 2, 1-3 days | 3, 1-2 days | 4, 3-4 days | 5, 5-6 days | 6, Every day (Higher score indicates increased vegetable consumption)
Time Frame: 3 months post-study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Comparison
Number analyzed (Participants) | 11 | 16
Participants | 9 | 5
Statistical Analysis 1: Comparison: Intervention vs Comparison; Test type: Superiority; p = 0.02, Regression, Logistic; Odds Ratio (OR) = 8.5, 95% CI 2-sided [1.3 to 54.6]

2. Primary Outcome: Count of Guardians Who Reported Being Confident or Very Confident That They Could Increase the Number of Vegetables the Child Eats Each Week
Description: Guardians who reported being Confident or Very Confident that they could increase the number of vegetables the child eats each week As measured by guardian self-efficacy and confidence questions related to modifiable lifestyle behaviors on a likert scale Question: How confident do you feel that you can increase the number of vegetables your child eats each week? Likert Scale: 1, Not confident = It is impossible for me to do this | 2, Somewhat confident = Maybe I can do this | 3, Confident = I think I can do this | 4, Very confident = I can absolutely do this (Higher score indicates better outcome than lower score on Likert scale)
Time Frame: 3 months post-study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Comparison
Number analyzed (Participants) | 11 | 16
Participants | 7 | 5
Statistical Analysis 1: Comparison: Intervention vs Comparison; Test type: Superiority; p = 0.015, Regression, Logistic; Odds Ratio (OR) = 9.98, 95% CI 2-sided [1.55 to 64.25]

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored over 3 months
Arm/Group | Intervention | Comparison
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/16
Other Adverse Events (participants affected / at risk) | 0/11 | 0/16

LIMITATIONS AND CAVEATS:
The study relied on self-reported measures of behaviors, which are subject to recall bias and social desirability bias and in addition we relied on reports from guardians about their child. The study had a relatively short follow-up period limiting our understanding of the long-term sustainability of intervention. The study sample was limited to a specific cultural group, which limits the generalizability of the findings to other cultural contexts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-31): https://cdn.clinicaltrials.gov/large-docs/57/NCT05419557/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-31): https://cdn.clinicaltrials.gov/large-docs/57/NCT05419557/ICF_001.pdf